CLINICAL TRIAL: NCT03535623
Title: Effects of Remote Ischemic Preconditioning During Free Flap Reconstruction in Head and Neck Cancer Patients With Preoperative Radiotherapy
Brief Title: RIPC During Free Flap With Preoperative Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Youn Joung Cho, MD, PhD, Clinical assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIPC during FF with RT
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Reperfusion Injury; Other Reconstructive Surgery; Radiotherapy
Keywords: remote ischemic preconditioning; free flap reconstruction; preoperative radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC (Experimental): Remote ischemic preconditioning (RIPC) consisted of 4 cycles of 5-min ischemia using pneumatic cuff pressure of 200 mmHg and 5-min reperfusion is applied to the upper arm of the patients in the RIPC group.
  Interventions: Other: remote ischemic preconditioning (RIPC)
- Sham-RIPC (Sham Comparator): Sham-RIPC consisted of 4 cycles of 5-min ischemia using pneumatic cuff pressure of < 10 mmHg and 5-min reperfusion is applied to the upper arm of the patients in the Sham-RIPC group.
  Interventions: Other: Sham-RIPC

INTERVENTIONS:
Other: remote ischemic preconditioning (RIPC) — RIPC consists of 4 cycles of 5-min ischemia using pneumatic cuff pressure of 200 mmHg and 5-min reperfusion.
  Arms: RIPC
Other: Sham-RIPC — Sham-RIPC consists of 4 cycles of 5-min ischemia using pneumatic cuff pressure of < 10 mmHg and 5-min reperfusion.
  Arms: Sham-RIPC

SUMMARY:
Remote ischemic preconditioning (RIPC) has shown organ-protective effects in many clinical settings including patients with ischemic heart disease. However its protective role in head and neck cancer patients with preoperative radiotherapy undergoing free flap reconstructive surgery has not yet been evaluated. The purpose of the current study is to evaluate the effect of RIPC on tissue oxygen saturation and skin temperature of the flap.

DETAILED DESCRIPTION:
Patients undergoing free flap reconstructive surgery for head and neck cancer with preoperative radiotherapy will be randomized to either remote ischemic preconditioning (RIPC) group or control group. On the day of surgery, after induction of anesthesia, RIPC, consisting of 4 cycles of 5-min ischemia (using pneumatic cuff pressure of 200 mmHg) followed by 5-min reperfusion at the upper arm, or sham-RIPC (pressure < 10 mmHg) will be induced in the RIPC or control group, respectively. Before completion of surgery, RIPC or sham-RIPC will be repeated. Tissue oxygen saturation and skin temperature of the flap will be recorded until postoperative day 1.

ELIGIBILITY:
Inclusion Criteria:

* Adult head and neck cancer patients undergoing free flap reconstructive surgery with preoperative radiotherapy

Exclusion Criteria:

* Radiotherapy within 4 weeks
* Body mass index < 18 kg/m^2 or > 35 kg/m^2
* Presence of AV fistula at the arm, any reason to protect arms
* Presence of vascular abnormality or discomfort at arms
* Peripheral vascular disease, peripheral neuropathy, or coagulopathy
* Uncontrolled diabetes mellitus
* Preoperative use of beta-blockers
* Refuse to enrol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
tissue oxygen saturation | postoperative day 1
  tissue oxygen saturation of the flap

SECONDARY OUTCOMES:
skin temperature | postoperative day 1
  skin temperature of the flap and the adjacent tissue

CONTACTS AND LOCATIONS:
Overall Officials: Youn Joung Cho, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided